CLINICAL TRIAL: NCT07177560
Title: Prospective Observational Study Assessing the Prophylactic Effect of Topical Diclofenac on Hand-Foot Syndrome in Patients With Colorectal and Gastric Cancer Receiving Capecitabine
Brief Title: Topical Diclofenac for Hand-Foot Syndrome Prevention in Colorectal and Gastric Cancer on Capecitabine (DICLO-HFS)
Acronym: DICLO-HFS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Principal Investigator, Department of Medical Oncology, Gazi University Faculty of Medicine, Gazi University
Other Study IDs: AESH-EKI-0022; 0022 (Other: Ankara Etlik City Hospital Ethics Committee)
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Gastric Cancer (GC); Capecitabine; Hand Foot Syndrome
Keywords: Hand-Foot Syndrome; Capecitabine; Topical Diclofenac; Chemotherapy Toxicity; Supportive Care
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Hand-Foot Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Topical Diclofenac: Patients with colorectal or gastric cancer receiving capecitabine who applied 1% topical diclofenac gel to the hands and feet twice daily throughout treatment. This group was managed according to physician preference and assessed weekly for the development of hand-foot syndrome (HFS).
- Observation: Patients with colorectal or gastric cancer receiving capecitabine who were actively monitored without prophylactic topical treatment. These patients were assessed weekly for the development of hand-foot syndrome (HFS).

SUMMARY:
Hand-foot syndrome (HFS) is a frequent adverse effect of capecitabine, presenting with redness, swelling, pain, and peeling of the skin on the palms and soles. These symptoms may impair daily activities and lead to treatment modifications.

This prospective observational study is being conducted at two tertiary oncology centers in Turkey to evaluate whether prophylactic use of topical diclofenac gel can prevent or delay the development of HFS in patients receiving capecitabine for colorectal or gastric cancer. Approximately 150 patients are enrolled and managed according to physician preference. Patients either receive topical diclofenac gel (applied twice daily to the hands and feet) or are followed with active monitoring.

The primary objective is to assess the incidence of grade 2 or 3 HFS. Secondary objectives include time to onset of HFS and the frequency of capecitabine dose reductions related to HFS.

DETAILED DESCRIPTION:
Hand-foot syndrome (HFS), also known as palmar-plantar erythrodysesthesia, is a common dermatologic toxicity of fluoropyrimidine chemotherapy such as capecitabine. Clinically significant HFS (grade ≥2) can negatively impact treatment adherence and quality of life by necessitating dose interruptions or reductions. The underlying mechanisms are not fully understood, but inflammatory pathways, including cyclooxygenase-2 (COX-2) signaling, are thought to contribute.

Preventive strategies for HFS remain limited. Celecoxib, a systemic COX-2 inhibitor, has been shown to reduce HFS incidence but is not widely adopted due to safety concerns. Topical diclofenac gel, a locally acting nonsteroidal anti-inflammatory drug (NSAID), represents a potential low-toxicity prophylactic approach.

This prospective, multicenter observational study is designed to evaluate the prophylactic effect of topical diclofenac in patients with colorectal or gastric cancer initiating capecitabine therapy. The study is conducted at Gazi University Faculty of Medicine and Ankara Etlik City Hospital. Eligible participants are adults scheduled to receive capecitabine-based therapy who have not received prior chemotherapy.

Participants are managed according to physician preference:

Topical diclofenac group: Patients apply 1% topical diclofenac gel to clean, dry skin on the hands and feet twice daily during capecitabine treatment.

Observation group: Patients are followed with active monitoring without prophylactic intervention.

The primary endpoint is the incidence of grade 2 or 3 HFS, assessed weekly using the Common Terminology Criteria for Adverse Events (CTCAE). Secondary endpoints include time to onset of HFS and the proportion of patients requiring capecitabine dose reductions due to HFS.

The planned enrollment is approximately 150 patients, with follow-up continuing until either the onset of clinically significant HFS or completion of capecitabine therapy.

ELIGIBILITY:
Inclusion Criteria

Age ≥18 years.

Histologically or cytologically confirmed colorectal or gastric cancer.

Planned capecitabine-based therapy (monotherapy or capecitabine plus oxaliplatin).

Planned starting capecitabine dose ≥2,000 mg/m²/day.

No prior systemic chemotherapy for the current malignancy.

Ability and willingness to attend weekly clinical assessments during treatment.

Written informed consent obtained.

Exclusion Criteria

Pre-existing dermatologic conditions affecting hands/feet (e.g., eczema, psoriasis) or peripheral neuropathy.

Sjögren's syndrome involving hands or feet.

Current or planned systemic NSAID use during capecitabine therapy.

Use of other HFS prophylaxis at baseline (e.g., topical NSAIDs other than diclofenac, pyridoxine).

Known hypersensitivity to diclofenac, aspirin, or other NSAIDs (e.g., history of asthma, urticaria, allergic reactions).

Planned initial capecitabine dose <2,000 mg/m²/day.

Anticipated inability to comply with weekly follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with histologically confirmed colorectal (colon or rectal) or gastric cancer who were initiating capecitabine-based therapy at two tertiary oncology centers in Ankara, Turkey (Gazi University; Ankara Etlik City Hospital). Patients were enrolled consecutively at treatment start and managed per treating physician practice into two observational cohorts: prophylactic 1% topical diclofenac gel vs active monitoring without prophylaxis. No prior systemic chemotherapy; weekly clinic assessments during therapy.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of grade ≥2 hand-foot syndrome (HFS) | Up to 24 weeks (from first capecitabine dose through study completion)
  Proportion of participants who develop grade ≥2 HFS during capecitabine therapy. HFS will be assessed weekly by oncology clinicians using the Common Terminology Criteria for Adverse Events (CTCAE). Numerator: participants with grade ≥2 HFS; Denominator: all enrolled participants.

SECONDARY OUTCOMES:
Time to onset of grade ≥2 hand-foot syndrome (HFS) | Up to 24 weeks (baseline to first event or end of study follow-up)
  Time (weeks) from the first capecitabine dose to the first documentation of grade ≥2 HFS per CTCAE. Participants without the event will be censored at end of treatment or end of follow-up.

OTHER OUTCOMES:
Treatment-emergent non-HFS adverse events (AEs) | Up to 24 weeks (from first capecitabine dose through study completion)
  Incidence and CTCAE grade of non-HFS AEs of interest (e.g., diarrhea, mucositis, neutropenia, thrombocytopenia). Reported as number (%) with any grade and grade ≥3 events.

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Ozdemir, MD, Study Chair — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Etlik City Hospital, Ankara
  - Gazi University, Ankara